CLINICAL TRIAL: NCT04780633
Title: The Effects of a PRECEDE-PROCEED Model-based Program on Genital Hygiene Behaviors: A Randomized Controlled Trial
Brief Title: PRECEDE-PROCEED Model-based Program on Genital Hygiene Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Manolya Parlas, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Approval No: 2017-3/20
Record Dates: First submitted 2021-02-21; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Genital Infection Female
Keywords: Genital hygiene behavior; Women's health; Precede-Proceed model; Health education; Nursing
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precede-Proceed based Training Program (Experimental): The experimental group is the group in which five training sessions interventions are applied.
  Interventions: Behavioral: Precede-Proceed based Training Program on Genital Hygiene Behaviors
- Control group (No Intervention): The control group is the group in which have no educational intervention.

INTERVENTIONS:
Behavioral: Precede-Proceed based Training Program on Genital Hygiene Behaviors — A Training Program for Genital Hygiene Behaviors prepared in line with the Precede-Proceed model was presented to the women in the experimental group. The trainings started one week after the pre-test data were collected and were conducted in a total of 5 sessions, each lasting an average of 40 minutes, once a week. At the end of the five-week training, a post-test was applied. In order to determine the behavior changes of the women in the experimental group, a follow-up test was applied 4 weeks after the training ended. At the end of the training, women were given a training booklet prepared by the researcher.
  Arms: Precede-Proceed based Training Program

SUMMARY:
The study was conducted to investigate the effect of a training program based on the PRECEDE-PROCEED Model on improving genital hygiene behaviors.It was carried out using experimental research design with pre-test and post-test, randomized and a control group. The study was conducted at Erzurum Saltuklu Family Health Center between June 2017 and January 2018. Of the women with genital infections, 120 women were included in the study, of which 60 were in the experimental group and 60 were in the control group. The data were collected by "Personal Information Form," "Genital Hygiene Knowledge, Attitude and Beliefs, Questionnaire" and "Genital Hygiene Behavior Inventory". In study, genital hygiene training intervention prepared according to the Precede-Proceed model was applied to the women in the experimental group. The women in the experimental group were measured at three different times: pre-test before training, post-test through training completition, and follow-up test after 4 weeks. The women in the control group did not receive any training intervention, the pre-test at the first encounter in the family health center and the post-test 5 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-49,
* married,
* At least primary school graduate,
* No mental and communication problems,
* No chronic disease,
* Non-pregnant.

Exclusion Criteria:

* Women who have entered menopause,
* Women who had received any training on genital hygiene before

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study was conducted women who diagnosed with genital infections.
Enrollment: 120 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
H1 hypothesis: PRECEDE-PROCEED training-based program affects on improving genital hygiene behavior. | 5 weeks
  Linear regression analysis was performed to determine the factors that are independently effective in determining the Genital Hygiene Behavior Inventory (GHBI) score differences between the pre-test and post-test measurements of the women in the experimental group.

CONTACTS AND LOCATIONS:
Locations (1):
- Manolya Parlas, Izmir, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No